CLINICAL TRIAL: NCT02637362
Title: Optimal Analgesia Following Metatarsal Surgery: A Prospective Randomised, Single-Blind Sham-Controlled Trial of Three Strategies
Brief Title: Optimal Analgesia for Forefoot Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Elizabeth Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr James Stimpson, Consultant Anaesthetist, Queen Elizabeth Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JSCP1
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Hallux Valgus; Conduction Block
MeSH Terms: conditions — Hallux Valgus; Heart Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ankle + Sham metatarsal (Active Comparator): Ankle block + sham metatarsal block
  Interventions: Procedure: Ankle block; Procedure: Sham metatarsal block
- Ankle + Metatarsal (Active Comparator): Ankle block + metatarsal block
  Interventions: Procedure: Ankle block; Procedure: Metatarsal block
- Metatarsal + sham ankle (Active Comparator): Metatarsal block + sham ankle block
  Interventions: Procedure: Sham ankle block; Procedure: Metatarsal block

INTERVENTIONS:
Procedure: Ankle block — Ultrasound guided ankle block of the tibial, superficial peroneal and deep peroneal nerves will be performed using a standardised technique
  Arms: Ankle + Metatarsal; Ankle + Sham metatarsal
Procedure: Sham ankle block — In the supine position with the hip and knee flexed, and the hip externally rotated, the skin from medial malleolus to Achilles tendon will be prepared with chlorhexidine 0.5% solution and allowed to dry. An ultrasound probe (linear array HFL25, Sonosite, Hitchin, UK) will be placed on a line from medial malleolus to achilles tendon to identify the posterior tibial artery and tibial nerve. A Stimuplex A50 needle (B-Braun) will be placed against the skin at the point at which the practitioner would normally have performed insertion of the needle. It will remain there for a total of 30 seconds and then will be removed.
  Arms: Metatarsal + sham ankle
Procedure: Metatarsal block — A metatarsal block will be performed using a standardised technique
  Arms: Ankle + Metatarsal; Metatarsal + sham ankle
Procedure: Sham metatarsal block — In the supine position, after the surgical incision has been sutured, a 25G standard bevel needle will be placed against the skin at the points at which the practitioner would normally have performed insertions of the needle. It will remain there for a total of 30 seconds and then be removed.
  Arms: Ankle + Sham metatarsal

SUMMARY:
A randomised trial comparing three analgesic strategies for patients undergoing forefoot surgery in a day-surgery setting.

DETAILED DESCRIPTION:
Forefoot surgery, including Scarf-Akin osteotomy surgery for bunion correction, is moderately painful orthopaedic surgery, commonly performed as a day-case procedure. Admission for opiate analgesia constitutes a failure of management and financial disadvantage to the healthcare organisation. The investigators seek to establish which technique will result in the best analgesia out of ankle block, metatarsal block, or a combination of the two. As analgesia constitutes part of a return to function, an additional aim is to determine whether either of these approaches will result in an objective functional benefit to the participants.

The trial seeks to recruit 23 patients into either of 3 groups: Ankle + sham metatarsal; sham Ankle + metatarsal; Ankle + Metatarsal.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, aged 18 years or above.
* Diagnosed with 1st metatarsal pathology requiring surgical correction
* Participant meets the criteria for operative management in our day-surgery unit

Exclusion Criteria:

* Contraindication to general anaesthesia
* Diabetic neuropathy affecting lower limbs
* Peripheral neuropathy affecting lower limbs of any aetiology
* Revision surgery
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Static pain score | 6 hours post-operatively
  Visual Analogue scores

SECONDARY OUTCOMES:
Dynamic pain scores | 6 hours post-operatively
  Visual Analogue scores
Dynamic pain scores | Day 1 post-operatively
  Visual Analogue scores
Dynamic pain scores | Day 7 post-operatively
  Visual Analogue scores
Assessment of functional recovery | 6 hours post-operatively
  Using Functional Recovery Index
Assessment of functional recovery | Day 1 post-operatively
  Using Functional Recovery Index
Assessment of functional recovery | Day 7 post-operatively
  Using Functional Recovery Index
Static pain score | Day 1 post-operatively
  Visual Analogue scores
Static pain score | Day 7 post-operatively
  Visual Analogue scores

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth Hospital NHS Trust, Kings Lynn, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No